CLINICAL TRIAL: NCT06602011
Title: Transcatheter Arterial Chemoembolization Combined With Lenvatinib Plus Tislelizumab for Intermediate-advanced Hepatocellular Carcinoma With Bile Duct Tumor Thrombus: A Multicenter, Single-arm, Real-world Study
Brief Title: Triple Therapy for Intermediate-advanced HCC With BDTT (TALENP002)
Status: Recruiting | Type: Observational
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Mao-Lin Yan, Department of Hepatobiliary Pancreatic Surgery, Fujian Provincial Hospital
Other Study IDs: TALENP002
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; bile duct tumor thrombus; TACE; Lenvatinib; Tislelizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Triple Therapy
  Interventions: Combination Product: TACE, Lenvatinib, combined with Tislelizumab group

INTERVENTIONS:
Combination Product: TACE, Lenvatinib, combined with Tislelizumab group — TACE, Lenvatinib [8mg(<60kg)/12mg(>60kg) orally daily] combination with Tislelizumab (200mg administered intravenous injection on Day 1 of each 21-day cycle). After the triple therapy, surgical resection is an option if assessed by the investigator to be feasible, or continued until disease progression or intolerable if not.

SUMMARY:
This is a multicenter, Single-arm, Real-world Study to evaluate the efficacy and safety of Transcatheter arterial chemoembolization (TACE), Lenvatinib combined with Tislelizumab (Triple Therapy) for patients with Hepatocellular Carcinoma (HCC) with bile duct tumor thrombus (BDTT).

DETAILED DESCRIPTION:
Surgical resection is considered to be the treatment of choice for Hepatocellular Carcinoma (HCC) combined with bile duct tumor thrombus (BDTT), but a significant proportion of patients with HCC combined with BDTT are unable to undergo surgical treatment at the time of initial diagnosis. For patients with unresectable advanced HCC combined with BDTT, conversion therapy is particularly important. Currently, there is relatively little literature related to the conversion treatment of HCC with BDTT. Several studies have confirmed that the transcatheter arterial chemoembolization (TACE), lenvatinib, combined with Tislelizumab (Triple Therapy) for the treatment of intermediate-advanced HCC can achieve better efficacy with an acceptable safety. However, there are no clinical studies or relevant literature reports on Triple Therapy for the treatment of HCC with BDTT. The present study is a multicenter, Single-arm, Real-world Study designed to evaluate the efficacy and safety of a triple therapy for the treatment of patients with HCC with BDTT.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years old;
2. Patients with clinical diagnosis of Hepatocellular Carcinoma (HCC) combined with bile duct tumor thrombus (BDTT) (refer to the diagnostic criteria of the Chinese Expert Consensus on Multidisciplinary Diagnosis and Treatment of HCC with BDTT (2020 Edition)), BCLC Stage B or Stage C, and unresectable HCC (decided after multidisciplinary discussion);
3. Patients who had not received any tumor-related targeted, immunotherapy, radiotherapy and chemotherapy before enrollment;
4. Patients with at least one measurable lesion according to the mRECIST criteria (measurable lesion with a CT/MRI scan length diameter ≥ 10 mm and measurable lesion has not received localized treatment such as TACE, radiofrequency, cryotherapy, etc.);
5. ECOG score: 0-1;
6. liver function Child-Pugh class A or B; if combined with obstructive jaundice, total bilirubin ≤50umol/L is required. If higher than 50umol/L, biliary drainage is recommended;
7. Blood routine: absolute neutrophil count ≥1.5×10^9/L, Hb≥8.5g/L, PLT≥75×10^9/L;
8. No history of severe cardiac arrhythmia or heart failure; no history of severe ventilatory dysfunction or severe pulmonary infection; no acute or chronic renal failure with creatinine clearance >40mL/min;
9. Expected survival time greater than 3 months.

Exclusion Criteria:

1. The tumor with extrahepatic metastasis or invaded adjacent organs;
2. Patients received other anti-tumor treatments;
3. Existence of contraindications to TACE;
4. History of allergy to the components or excipients of Lenvatinib or Tislelizumab;
5. The patient has any active autoimmune disease or has an autoimmune disease with expected relapse. Patients are on immunosuppressive or systemic hormone therapy for immunosuppression;
6. Patients with proteinuria suggestive of ≥ 1 + in routine urine will undergo a 24-hour urine protein test for patients with ≥ 1 g of 24-hour urine protein;
7. Patients with co-morbidities of other malignant tumors;
8. Patients with co-morbid psychiatric disorders;
9. Patients with pregnant or lactating women;
10. Patients with organ transplant patients;
11. Patients with hypothyroidism or hyperthyroidism.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intermediate-advanced Hepatocellular Carcinoma With Bile Duct Tumor Thrombus
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate, ORR | Four weeks after the initiation of medication until the day before surgery
  The Objective response rate (ORR) was defined as the complete response (CR) rate or the partial response (PR) rate according to mRECIST.

SECONDARY OUTCOMES:
Overall survival, OS | From date of enrollment until the date of death from any cause, assessed up to 60 months
  The Overall survival (OS) was defined as the time between receiving treatment and observing death or loss of follow-up for any reason.
Progression free survival, PFS | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  The Progression free survival (PFS) was defined as the time between the start of treatment and the progression of intrahepatic and/or extrahepatic tumors, or the occurrence of death or loss of follow-up for any reason.
The Disease control rate, DCR | Four weeks after the initiation of medication until the day before surgery
  The Disease control rate (DCR) was defined as the complete response (CR) rate or the partial response (PR) rate or stable disease (SD) rate according to mRECIST.
Conversion resection rate, CRR | Four weeks after the initiation of medication until the day before surgery
  The Conversion resection rate (CRR) was defined as the patient who reach the resectable criterion after treatment and accepted operation.
Toxicity Adverse events | From the initiation of medication, with recordings made whenever an adverse reaction occurs, assessed up to 12 months
  Grade 1-5 AEs according to NCI-CTCAE V5.0.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Zhongshan Hospital of Xiamen University, Xiamen, Fujian
  - First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhangzhou Affiliated Hospital of Fujian Medical University, Zhangzhou, Fujian

IPD SHARING:
Plan to Share IPD: No